CLINICAL TRIAL: NCT03831542
Title: Follicular Flushing in Patients With Mono-follicular Growth
Brief Title: Effect of Follicular Flushing in Patients With Mono-follicular Growth Undergoing In Vitro Fertilization
Status: Completed | Type: Observational
Sponsor: Centrum Clinic IVF Center (Other)
Responsible Party: Principal Investigator, Emre Göksan Pabuçcu, Emre G. Pabuccu, Assoc. Prof., Centrum Clinic IVF Center
Other Study IDs: 1
Record Dates: First submitted 2019-02-02; First posted 2019-02-06 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Invitro Fertilization; Diminished Ovarian Reserve; Oocyte
Keywords: follicular flushing; double lumen needle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- direct aspiration group: Transvaginal ultrasound-guided oocyte retrieval was performed 36 hours after ovulation trigger. A 17-gauge double lumen needle will be used to aspirate a single follicle without flushing. If an oocyte is obtained, the subject will be assigned to group 1. If not, operator will proceed with follicular flushing.
  Interventions: Behavioral: direct follicular aspiration
- flushing group: If an oocyte is not obtained with direct aspiration, operator will proceed to follicular flushing and the subject will be assigned to group 2 if an oocyte is obtained following follicular flushing.
  Interventions: Behavioral: follicular flushing

INTERVENTIONS:
Behavioral: direct follicular aspiration — direct follicular aspiration
  Groups: direct aspiration group
Behavioral: follicular flushing — follicular flushing
  Groups: flushing group

SUMMARY:
Retrieval of an oocyte from a follicle relies on the release of the cumulus-oocyte-complex (COC) from the follicular wall into the lumen, thereby allowing aspiration by a needle. Flushing the follicle with multiple aspirations from the same follicle is used as a means to increase the ratio of COC per aspirated follicle. Data showed that follicular flushing is not superior to direct aspiration either in normally responding patients or in poor responders undergoing in vitro fertilization (IVF). There is no data in the literature regarding the issue in patients with mono-follicular growth. Direct aspiration or repeatedly flushing the follicle for those with a single follicle will be investigated.

DETAILED DESCRIPTION:
Oocyte retrieval procedure This study aims to evaluate the effect of follicular flushing during oocyte retrieval procedure in patients with only one follicle. Double lumen needle will be used and direct follicular aspiration without flushing will be performed for all patients. If an oocyte will be obtained, the patient will be assigned to group A. If not, at least 1 course of follicular flushing will be used until retrieval of an oocyte and the patient will be assigned to group B.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-40 years
* primary infertility
* diminished ovarian reserve with single mature follicle on the day of oocyte retrieval

Exclusion Criteria:

* natural cycle IVF
* presence of endometriosis/endometrioma(s)
* Absence of cumulus oocyte complex following oocyte retrieval
* Severe male factor infertility
* Pre-implantation genetic screening cycles

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women undergoing oocyte retrieval procedure due to primary infertility
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
mature oocyte | during oocyte retrieval procedure
  Confirmation of cumulus oocyte complex (COC) after microscopic examination of follicular fluid by a senior embryologist for each patient.

SECONDARY OUTCOMES:
fertilization rate after micro-injection | 24 hours after microinjection procedure
  Confirmation of pronuclei formation on the following day of microinjection by a senior embryologist in each patient.
clinical pregnancy rate per embryo transfer | untill 6 weeks
  Confirmation of fetal cardiac activity on 5th or 6th week of gestation by a senior obstetrician in each pregnancy case.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Pabuccu, MD, Study Director — Centrum Clinic IVF Center
Locations (1):
- Centrum Clinic IVF Center, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] von Horn K, Depenbusch M, Schultze-Mosgau A, Griesinger G. Randomized, open trial comparing a modified double-lumen needle follicular flushing system with a single-lumen aspiration needle in IVF patients with poor ovarian response. Hum Reprod. 2017 Apr 1;32(4):832-835. doi: 10.1093/humrep/dex019. PMID 28333185
- [Result] Haydardedeoglu B, Gjemalaj F, Aytac PC, Kilicdag EB. Direct aspiration versus follicular flushing in poor responders undergoing intracytoplasmic sperm injection: a randomised controlled trial. BJOG. 2017 Jul;124(8):1190-1196. doi: 10.1111/1471-0528.14629. Epub 2017 May 2. PMID 28276148